CLINICAL TRIAL: NCT02940210
Title: A Randomized, Single-blind, Multi-center, Phase III Clinical Trail to Evaluate the Efficacy and Safety of Adhesion Barrier Mediclore Versus no Treatment in Patients With Total Thyroidectomy
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Adhesion Barrier Mediclore Versus no Treatment in Patients With Total Thyroidectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CGBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CG-AHS004
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Patients With Thyroidectomy (Scheduled)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediclore® (Experimental): adhesion barrier Mediclore 5cc, to apply medical device fully around thyroid gland following thyroidectomy
  Interventions: Device: Mediclore® (adhesion barrier)
- No treatment (No Intervention): No treatment, standard treatment for thyroidectomy

INTERVENTIONS:
Device: Mediclore® (adhesion barrier)
  Arms: Mediclore®

SUMMARY:
A randomized, single-blind, multi-center, Phase III clinical trial to evaluate the efficacy and safety of adhesion barrier Mediclore versus no treatment in patients with total thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female at least 20 years of age
* Patients without clinically significant lab
* Patients scheduled for thyroidectomy

Exclusion Criteria:

* Another clinical trials within 1 month
* History of previous surgery on same position
* Anticoagulant, general steroids within a week from surgery
* Immunosuppression or autoimmune disease
* General or local infection
* Serious diseases (heart failure, renal failure, liver failure, uncontrolled hypertension, diabetes mellitus, coagulation deficiencies)
* Incompatible medications
* History of drug or alcohol abuse, mental disorder
* Pregnant or lactating women and fertile women who is not using proper contraceptive method
* History of esophagus diseases
* Keloid symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Adhesion incidence rate following 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No